CLINICAL TRIAL: NCT04418622
Title: Evolution of the Endonasal Microbiota After Endoscopic and Local Treatment or Local Treatment Alone in Patients With Chronic Rhinosinusitis
Brief Title: Evolution of the Endonasal Microbiota in Patients With Chronic Rhinosinusitis
Acronym: METEL-RC
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: METEL-RC (29BRC19.0162)
Record Dates: First submitted 2020-06-04; First posted 2020-06-05 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Chronic Sinusitis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective

SUMMARY:
Chronic rhinosinusitis (CRS) is defined according to the French society of otorhinolaryngology as chronic non-mechanical damage to the nasal structures, excluding infectious damage to the sinus structures. The duration of the chronic impairment must be at least 12 consecutive weeks. It causes many symptoms such as rhinorrhea, nasal blockage and anosmia. It is a poorly understood pathology that affects a large part of the population. Its prevalence has increased significantly over the past 30 years. It affects about 11% of the population in Europe. It has become one of ten high-cost medical conditions for employers. Initially, it was accepted that CRS was due to chronic nasal infection. It is very debilitating for patients leading to a major consultation with practitioners (general practitioners and ENT specialists). Many treatments are used such as nose washes, nasal or oral corticosteroids, antibiotic therapy or even surgical management is possible. Thèses treatments allow an improvement in the symptomatology but no treatment allows a stable result over time, making long-term treatments essential.

Today, it is recognized that CRS has a multifactorial etiology including inflammatory processes, hyperresponsiveness of the nasal mucosa and abnormalities in immune phenomena. The endonasal microbiota plays a role in these processes. Germs like Staphylococcus aureus and Pseudomonas aeruginosa were identified as pathogens in CRS in the first studies with bacterial cultures. Thanks to the 16S ribosomal RNA sequencing technique, recent studies have demonstrated a modification in the diversity and abundance of the microbiota in patients with CRS compared to healthy subjects, notably with a modification of the germs of the firmicutes group. .

Few studies have studied the modification of the microbiota with the treatment of CRS today. However, local treatments based on nosewashing with physiological saline associated with local corticosteroids and endoscopic treatments lead to an improvement in the symptomatology for patients suffering from CRS. This study will describe the modification of endonasal microbiota in différent conditions, such medical and surgical treatments, that usually improve patients symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* patients without chronic rhinosinusitis who undergo a nasal surgery
* patients with chronic rhinosinusitis who undergo a medical or surgical treatment

Exclusion Criteria:

* minor patients
* pregnant or lactating women
* patients undergoing antibiotic therapy in the month preceding the start of the study
* patients with immunosuppression
* ENT cancer or other cancer in progress
* primary ciliary dyskinesia or cystic fibrosis
* Systemic vasculitis (Wegener, Gougerot-Sjögren ...)
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients without chronic rhinosinusitis who undergo a nasal surgery and patients with chronic rhinosinusitis who undergo a medical or surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
description of biodiversity of the microbiota | six month
  Shannon index
richness of samples | six month
  number of OTU (operational taxonomic unit)

SECONDARY OUTCOMES:
patient quality of life | six month
  specific questionnaire Sino-nasal Outcome Test (SNOT-22). minimum 0 maximum 110. The higher the score the greater the impact of the symptoms on quality of life.
rhinosinusal inflammation | six month
  lund kennedy score. Minimum 0. maximum 10. the higher the score the greater the signs of chronic rhinosinusitis.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending five years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the international committee of Brest UH. Requestors will be required to sign and complete a data access agreement.